CLINICAL TRIAL: NCT00146146
Title: Role of Testosterone and Its Metabolites Regarding Different Physiological Functions in Subjects Affected by Gender Identity Disorder (FtM Transsexuals)
Brief Title: Testosterone and Its Metabolites in GID
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Unita Complessa di Ostetricia e Ginecologia (Other)
Collaborators: Schering-Plough (Industry)
Responsible Party: Dr Meriggiola Maria Cristina, Unita Complessa di Ostetricia e Ginecologia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GID/2004
Record Dates: First submitted 2005-09-01; First posted 2005-09-05 (Estimated); Last update posted 2018-03-21 (Actual); Status verified 2009-02

CONDITIONS: Transsexualism
Keywords: transsexualism; testosterone; dihydrotestosterone; estradiol
MeSH Terms: conditions — Transsexualism | interventions — testosterone undecanoate; Letrozole; Dutasteride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: testosterone undecanoate alone — 1000 mg/12 weeks
  Other Names: Nebid
Drug: testosterone undecanoate plus letrozole — TU 1000 mg/12 weeks Letrozole 2.5 mg/day
  Other Names: Nebid
Drug: testosterone undecanoate plus dutasteride — TU 1000 mg/12weeks Dutasteride 0.5 mg/day
  Other Names: Nebid; Avodart

SUMMARY:
The purposes of this study are:

* to determine the role of testosterone versus dihydrotestosterone with respect to the following physiological functions: bone metabolism, body composition, insulin resistance and lipid profile
* to determine the role of testosterone and dihydrotestosterone versus estradiol with respect to the following physiological functions: bone metabolism, body composition, insulin resistance and lipid profile

DETAILED DESCRIPTION:
BACKGROUND GID is a psychic disorder in which an otherwise normal person feels like he/she is a member of the opposite sex to which she/he belongs biologically. These patients require hormonal treatment to suppress the somatic characteristics of their own sex and to develop the somatic characteristics of the other sex. After psychotherapy and a period of hormonal treatment, they undergo surgical sex reassignment which, in the case of FtM subjects, consists of hystero-adnexectomy, reductive mastoplasty and possibly penile reconstruction. Thereafter, and for their entire life, they must be treated with testosterone (T) to maintain androgen-dependent physiological functions.

RATIONALE After sex-reassignment surgery, FtM subjects must be treated with T for their entire life in order to maintain androgen-estrogen dependent physiological functions.

These subjects represent an interesting model for the study of the effects of testosterone and its metabolites on different physiological functions. As of now, there is no information that the androgen receptors differ in males and females. Therefore, induction of the androgen effects in the FtM subjects can be considered similar to those in hypogonadal men and FtM subjects can serve as a model of the hypogonadal male.

Therefore, the aim of this trial is to evaluate the effects of selective steroid replacement on different physiological functions. In particular in this study we will evaluate the relative role of testosterone, DHT and estradiol on the different physiological functions. For these purposes, we will administer testosterone undecanoate alone (Group A) or in combination with letrozole, an aromatase inhibitor (Group B). A third group of FtM subjects will be treated with TU plus dutasteride (Group C).

In view of the development of selective androgen receptor modulators, the understanding of the relative role of each steroid on different physiological functions will provide useful information for future therapeutic indications. The information collected in this study will greatly help to optimize the long-term treatment of FtM subjects.

In particular, in this study, we will test the following questions:

* what is the role of testosterone vs. DHT on the physiological functions evaluated in this study i.e. bone metabolism, body composition, insulin resistance and lipid profile (Group B vs. Group C)
* what is the role of testosterone and DHT vs estradiol on the physiological functions evaluated in this study i.e. bone metabolism, body composition, insulin resistance and lipid profile (Group C vs. Group A)

DESIGN

For this purpose, in this study we will treat FtM castrated, subjects for 54 weeks with:

* testosterone undecanoate 1000 mg 6-12 weeks (injection at week 0, 6, 18, 30, 42 and 54)(n=5) (Group A)
* testosterone undecanoate 1000 mg 6-12 weeks (injection at week 0, 6, 18, 30, 42 and 54) mg/day plus letrozole 2.5 mg/day (n=5) (Group B)
* testosterone undecanoate 1000 mg 6-12 weeks (injection at week 0, 6, 18, 30, 42 and 54) plus dutasteride 0.5 mg/day (n=5) (Group C)

Overall study design and plan-description Prospective, phase III, randomized study design will be used. The study consists of a control phase lasting 3 weeks and a 54-week treatment period.

Control phase: (will last 3 weeks: In this period, subjects will provide three fasting (at least 10 hours) blood samples and one urine sample. Subjects will undergo 2 visits to ensure fulfillment of inclusion criteria and, absence of exclusion criteria, to determine state of health and to be informed about the purposes of the study. During the two visits, they will undergo:

* blood drawings for measurements of: LH, FSH, estradiol, testosterone DHEAS, total cholesterol, HDL cholesterol, triglycerides, insulin, glucose, leptin, adiponectin, uric acid, urea, creatinine, Na, K, Ca, P, Mg, Cl, total protein, bone alkaline phosphate, PTH, osteocalcin, crosslaps, 25(OH) vit D, H RANKL, osteoprotegerin.
* anthropometry: weight, measures
* DEXA for bone mass determination and body composition
* physical examination
* a sexual and behavioral questionnaire
* a pain questionnaire

Treatment phase All injections will be administered by the investigator or co-investigators for the entire study. Fasting (10 hours) blood samples will be taken (immediately before giving the injections) every time subjects come for injections (week 0, 6, 18, 30 and 42) and at the end of the treatment phase. On these occasions, a physical examination including weight, blood pressure and pulse rate checks will be performed. Volunteers will be asked to complete a sexual and behavioral questionnaire and a pain questionnaire during these visits.

At week 6, 18, 30 and 42 the following tests will be performed:

* blood drawings for measurements of: LH, FSH, estradiol, testosterone, DHT, total cholesterol, HDL cholesterol, triglycerides, insulin, glucose, leptin, adiponectin, uric acid, urea, creatinine, Na, K, Ca, P, Mg, Cl, total protein.
* anthropometry: weight, measures
* physical examination
* sexual and behavioral questionnaire
* pain questionnaire

At week 54 the following tests will be performed:

* blood drawings for measurements of: LH, FSH, estradiol, testosterone, DHT, DHEAS, total cholesterol, HDL cholesterol, triglycerides, insulin, glucose, leptin, adiponectin, uric acid, urea, creatinine, Na, K, Ca, P, Mg, Cl, total protein, bone alkaline phosphate, PTH, osteocalcin, crosslaps, 25(OH) vit D, H RANKL, osteoprotegerin.
* anthropometry: weight, measures
* DEXA for bone mass determination and body composition
* physical examination
* sexual and behavioral questionnaire
* pain questionnaire

Measurements:

Blood samples(10 hours from last food intake). Blood collections will be carried out by venipuncture. After resting at room temperature for 30 min, the sample will be centrifuged at 3000 rpm for 10 min. Serum samples (about 10 ml) from each blood sample will be stored at -20°C for analysis.

Physical examinations:

They will include inspection of external genitalia (clitorides) and a visit to detect appearance of acne and gynecomastia.

Sexual function and behavior questionnaire:

In the sexual and behavior questionnaire the subjects will judge their sexual activity and behavior in the period between visits. The subjects have the possibility to making additional comments about important events and disturbances.

SELECTION OF STUDY POPULATION:

Healthy female FtM subjects, who have undergone SR surgery (hystero-adnexectomy) will be recruited to participate in this study. Healthy female subjects between 18 to 45 years of age will be enrolled in the study according to Inclusion/Exclusion Criteria listed below. They will be informed about the nature, aim and objectives of the study and will be required to give their written consent to participate in the study. The presence of the inclusion criteria and the absence of the exclusion criteria will be documented in the Case Report Forms (CRF).

ELIGIBILITY:
Inclusion Criteria:

Healthy biological females, between 18 and 45 years of age:

* SR surgery performed
* Body Mass Index (BMI) between 20 and 29 kg/m²; (body weight in kilograms divided by body height in meters squared)
* Clinical examination without pathological findings relevant to the study
* Clinico-chemical laboratory values do not suggest an illness
* Written Consent Form has been signed
* High probability of a good compliance and termination of the study

Exclusion Criteria:

Subjects cannot be enrolled in this study if one or more of the following criteria apply:

* Participation in another clinical trial within the 30 days preceding the first administration
* Simultaneous participation in another clinical trial
* Subjects institutionalized or imprisoned by order of the court
* Subject who compete in sports which use IOC drug monitoring
* Serious organic or psychic disease suspected from history and/or clinical examination
* Diseases (especially tumors) that might represent an actual contraindication for testosterone
* Past or present history of thrombotic or embolic diseases
* Hypertension requiring therapy (BP 140/90 mmHg)
* Diabetes mellitus requiring therapy
* Acute or chronic hepatic diseases
* Manifest renal diseases with renal dysfunction
* Severe internal diseases as well as use of any medication to treat such
* Biochemical and/or hematological laboratory values beyond normal ranges unless the Investigator confirms that the deviations are of no clinical relevance
* Any indication of chronic use of drugs, alcohol, opiates or recreational drugs
* Use of any drug known to affect biotransformation of testosterone and/or progestin, e.g. chlorcycline, phenobarbital, phenylbutazone, aminophenazone within the 30 days preceding the first administration of the test medication and during the study
* Use of oral anticoagulatory drugs within the 30 days preceding the first administration of the test medication and during the study
* Any oral or transdermal hormone medication within the 12 weeks preceding the first administration and during the study
* Probability of poor compliance and termination of the study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2005-05; Primary Completion 2006-05 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
bone metabolism | baseline and end of the study
insulin resistance | baseline and end of the study
lipid profile | baseline and end of the study

SECONDARY OUTCOMES:
sexual function | baseline and end of the study
mood | baseline and end of the study
pain | baseline and end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Cristina M Meriggiola, MD, Principal Investigator — University of Bologna
Locations (1):
- Clinic of Obstetrics and Gynecology - S. Orsola Hospital, Bologna, Italy

REFERENCES:
- [Background] Cherrier MM, Matsumoto AM, Amory JK, Ahmed S, Bremner W, Peskind ER, Raskind MA, Johnson M, Craft S. The role of aromatization in testosterone supplementation: effects on cognition in older men. Neurology. 2005 Jan 25;64(2):290-6. doi: 10.1212/01.WNL.0000149639.25136.CA. PMID 15668427
- [Background] Reddy DS. Testosterone modulation of seizure susceptibility is mediated by neurosteroids 3alpha-androstanediol and 17beta-estradiol. Neuroscience. 2004;129(1):195-207. doi: 10.1016/j.neuroscience.2004.08.002. PMID 15489042
- [Background] Swaab DF. Sexual differentiation of the human brain: relevance for gender identity, transsexualism and sexual orientation. Gynecol Endocrinol. 2004 Dec;19(6):301-12. doi: 10.1080/09513590400018231. PMID 15724806
- [Background] Turner A, Chen TC, Barber TW, Malabanan AO, Holick MF, Tangpricha V. Testosterone increases bone mineral density in female-to-male transsexuals: a case series of 15 subjects. Clin Endocrinol (Oxf). 2004 Nov;61(5):560-6. doi: 10.1111/j.1365-2265.2004.02125.x. PMID 15521957
- [Background] Cherrier MM, Anawalt BD, Herbst KL, Amory JK, Craft S, Matsumoto AM, Bremner WJ. Cognitive effects of short-term manipulation of serum sex steroids in healthy young men. J Clin Endocrinol Metab. 2002 Jul;87(7):3090-6. doi: 10.1210/jcem.87.7.8570. PMID 12107206
- [Background] Bagatell CJ, Heiman JR, Rivier JE, Bremner WJ. Effects of endogenous testosterone and estradiol on sexual behavior in normal young men. J Clin Endocrinol Metab. 1994 Mar;78(3):711-6. doi: 10.1210/jcem.78.3.8126146.
- [Background] Amory JK, Watts NB, Easley KA, Sutton PR, Anawalt BD, Matsumoto AM, Bremner WJ, Tenover JL. Exogenous testosterone or testosterone with finasteride increases bone mineral density in older men with low serum testosterone. J Clin Endocrinol Metab. 2004 Feb;89(2):503-10. doi: 10.1210/jc.2003-031110. PMID 14764753
- [Background] Levy A, Crown A, Reid R. Endocrine intervention for transsexuals. Clin Endocrinol (Oxf). 2003 Oct;59(4):409-18. doi: 10.1046/j.1365-2265.2003.01821.x. No abstract available. PMID 14510900
- [Background] Tangpricha V, Ducharme SH, Barber TW, Chipkin SR. Endocrinologic treatment of gender identity disorders. Endocr Pract. 2003 Jan-Feb;9(1):12-21. doi: 10.4158/EP.9.1.12. PMID 12917087
- [Background] Moore E, Wisniewski A, Dobs A. Endocrine treatment of transsexual people: a review of treatment regimens, outcomes, and adverse effects. J Clin Endocrinol Metab. 2003 Aug;88(8):3467-73. doi: 10.1210/jc.2002-021967. PMID 12915619